CLINICAL TRIAL: NCT00956943
Title: Assessment of High Dose Transdermal Nicotine for Fast Metabolizers of Nicotine
Acronym: HDP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Robert Schnoll, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 809716; R21DA026889 (NIH)
Record Dates: First submitted 2009-07-23; First posted 2009-08-11 (Estimated); Results first posted 2013-03-18 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Nicotine Dependence
Keywords: nicotine dependence; nicotine replacement therapy; transdermal nicotine; nicotine metabolism; high dose
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 21mg transdermal nicotine + placebo patch (Active Comparator): 21mg transdermal nicotine + placebo patch
  Interventions: Drug: Nicoderm CQ transdermal nicotine; Drug: placebo
- 42mg transdermal nicotine (Experimental): 42mg transdermal nicotine
  Interventions: Drug: Nicoderm CQ transdermal nicotine

INTERVENTIONS:
Drug: Nicoderm CQ transdermal nicotine — Transdermal nicotine patch (21mg vs. 42mg), 8 weeks
Drug: placebo — placebo patch
  Arms: 21mg transdermal nicotine + placebo patch

SUMMARY:
Unfortunately, the investigators still need to assess and identify novel ways to help people quit smoking. Differences between people in terms of how fast they metabolize nicotine influences response to transdermal nicotine patches, the most popular nicotine dependence treatment, and it affects plasma levels of nicotine from treatment. These studies suggest that fast metabolizers of nicotine may show better quit rates if they receive higher doses of transdermal nicotine. This preliminary study is designed to assess, for the first time, whether fast nicotine metabolizers show higher quit rates if given high dose transdermal nicotine, versus standard dose. The study findings may help to support a subsequent large trial to assess standard versus high dose transdermal nicotine for slow versus fast metabolizers of nicotine, which may lead to a more personalized approach to treating nicotine dependence using the nicotine patch to improve therapeutic benefits of transdermal nicotine.

DETAILED DESCRIPTION:
Novel approaches to treating nicotine dependence remain a priority. The transdermal nicotine patch is the most widely used form of tobacco dependence treatment, but only ~1 in 5 smokers who use this treatment achieve cessation. One factor that may contribute to a poor response to transdermal nicotine is inter-individual variability in the rate of nicotine metabolism, which can be measured in saliva by the ratio of 3'hydroxycotinine (3-HC) to its precursor cotinine.

Two clinical trials with transdermal nicotine have shown that the 3-HC/cotinine ratio predicts response to transdermal nicotine such that faster metabolizers of nicotine (higher 3-HC/cotinine ratios) have lower quit rates, vs. slower nicotine metabolizers. Among abstainers in these trials, the 3-HC/cotinine ratio also predicts therapeutic levels of nicotine on transdermal nicotine, with faster metabolizers of nicotine exhibiting lower nicotine. Thus, faster metabolizers of nicotine may require higher nicotine doses to achieve the same therapeutic benefit from transdermal nicotine as do slow nicotine metabolizers.

To date, clinical trials have shown that, compared to the standard dose of transdermal nicotine (21mg), higher doses (42mg) have no significant effect on quit rates. However, no trial of high dose transdermal nicotine considered inter-individual variability in the rate of nicotine metabolism. Thus, as a preliminary step toward conducting a fully-powered, randomized clinical trial to assess standard vs. high dose transdermal nicotine for slow vs. fast metabolizers of nicotine, we propose to evaluate, for the first time, the efficacy of high-dose transdermal nicotine (vs. standard dose) among fast metabolizers of nicotine (i.e., upper quartile of the 3-HC/cotinine ratio distribution).

We chose only fast metabolizers of nicotine for this trial since: 1) slow metabolizers of nicotine exhibit high quit rates on standard transdermal nicotine and may experience adverse effects from higher doses; and 2) as a "proof of concept" R21 application, our primary objective is to test whether high doses of nicotine increase quit rates among fast metabolizers of nicotine. Specifically, smokers who are fast metabolizers of nicotine will receive counseling and will be randomized to: 1) standard (1 X 21mg patch and 1 X placebo patch), or 2) high dose (2 x 21mg patches) transdermal nicotine.

The primary outcome is biochemically-verified 7-day point prevalence cessation after 8 weeks of treatment. Differences in patch-related side effects and mediators of transdermal nicotine effects (e.g., nicotine levels, withdrawal) across the study conditions will also be assessed.

Ultimately, this line of research hopes to provide the evidence necessary to translate research on the 3-HC/cotinine ratio to clinical practice for the treatment of tobacco dependence. Specifically, this research may show that a measure of nicotine metabolism rate could be used to maximize the therapeutic benefits of transdermal nicotine by providing slow metabolizers of nicotine with a standard patch dose and fast metabolizers of nicotine with high dose transdermal nicotine. Identifying an effective treatment for faster metabolizers of nicotine is also critical since these individuals are at increased risk for lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 18-45 who smoke > 10 cigarettes/ day;
2. Able to communicate in English;
3. Able to use NRT safely (e.g., no allergy to latex);
4. Able to provide written informed consent for study procedures;
5. Residing in the geographic area for at least 6 months; and
6. A 3-HC/cotinine ratio in the top quartile of the distribution (Schnoll et al., 2008). Age 45 was selected as an upper limit to reduce the likelihood of adverse effects from high dose transdermal nicotine.

Exclusion Criteria:

1. History of substance abuse or currently receiving treatment for substance abuse (e.g., alcohol, opioids, cocaine, marijuana);
2. Current (last 6-months) alcohol consumption that exceeds 25 standard drinks/week.
3. Current use or discontinuation within last 14 days of:

   * Smoking cessation medications (bupropion, Chantix, NRT);
   * Antipsychotics, atypicals, mood-stabilizers, anti-depressants (tricyclics, SSRIs, MAOIs), anti-panic agents, anti-obsessive agents, anti-anxiety agents, stimulants);
   * Medication for pain;
   * Anti-coagulants;
   * Heart medications;
   * Daily medication for asthma or diabetes.
4. Women who are pregnant, planning a pregnancy, or lactating;
5. History or current diagnosis of psychosis, major depression or bipolar disorder, psychotic disorder, or generalized anxiety disorder;
6. Serious/unstable disease within the past 6 months (e.g., cancer [but melanoma], HIV/AIDS);
7. History of epilepsy or seizure disorder;
8. History or diagnosis within the last 6 months of abnormal rhythms and/or tachycardia (>100 beats/minute); history or current diagnosis of COPD, cardiovascular disease (stroke, angina), heart attack in the last 6 months, uncontrolled hypertension (SBP>150 or DBP>90);
9. History of kidney or liver failure.
10. Any medical condition or medication that could compromise safety as determined by a study physician;
11. Inability to provide informed consent or complete the study tasks as determined by the Principal Investigator or study physician.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Schnoll, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Media ads asked treatment-seeking smokers to call for information about a smoking cessation program and to have their initial eligibility reviewed. Participants interested in the clinical trial and initially eligible attended an in-person session to determine their final eligibility. Recruitment was from 2009-2011.
Pre-assignment Details: To be eligible, participants had to be: between age 18 and 55, smoke >10 cigarettes/day, and able to communicate in English. In addition, participants had to have a 3-HC/cotinine ratio that placed them in the top 3 quartiles of the 3-HC/cotinine ratio distribution to be consider fast nicotine metabolizers, which was >.18.
Groups:
- 21mg Transdermal Nicotine + Placebo Patch: 21mg transdermal nicotine + placebo patch
  Nicoderm CQ transdermal nicotine : Transdermal nicotine patch (21mg vs. 42mg), 8 weeks
  placebo : placebo patch
- 42mg Transdermal Nicotine: 42mg transdermal nicotine
  Nicoderm CQ transdermal nicotine : Transdermal nicotine patch (21mg vs. 42mg), 8 weeks
Period: Overall Study
Arm/Group | 21mg Transdermal Nicotine + Placebo Patch | 42mg Transdermal Nicotine
Started | 43 | 44
Baseline | 43 | 44
Completed | 34 | 34
Not Completed | 9 | 10
Not completed — Lost to Follow-up | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 21mg Transdermal Nicotine + Placebo Patch | 42mg Transdermal Nicotine | Total
Number analyzed (Participants) | 43 | 44 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 44 | 87
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (9.0) | 38.8 (9.0) | 38 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 21 | 21 | 42
Region of Enrollment [Number; unit: participants]
  United States | 43 | 44 | 87

OUTCOME MEASURES:

1. Primary Outcome: Biochemically Verified 7-day Point Prevalence Abstinence at the End of 8 Weeks of Treatment
Description: quit rate verified with carbon monoxide breath sample (abstinence: less than or equal to 10ppm)
Time Frame: After 8 weeks of treatment with the patch, outcome will be measured.
Population: intent to treat
Measure: Number; unit: participants
Arm/Group | 21mg Transdermal Nicotine + Placebo Patch | 42mg Transdermal Nicotine
Number analyzed (Participants) | 43 | 44
participants | 10 | 13

2. Secondary Outcome: Side Effects
Description: frequency of serious adverse events
Time Frame: 8 weeks
Population: intent to treat
Measure: Number; unit: events
Arm/Group | 21mg Transdermal Nicotine + Placebo Patch | 42mg Transdermal Nicotine
Number analyzed (Participants) | 43 | 44
events | 0 | 1

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | 21mg Transdermal Nicotine + Placebo Patch | 42mg Transdermal Nicotine
Serious Adverse Events (participants affected / at risk) | 0/43 | 1/44
Other Adverse Events (participants affected / at risk) | 0/43 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 21mg Transdermal Nicotine + Placebo Patch (N=43) | 42mg Transdermal Nicotine (N=44)
influenza (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a proof of concept trial and, as such, was inadequately powered to detect statistically significant treatment arm effects and did not include a long-term follow-up assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes